CLINICAL TRIAL: NCT04045769
Title: A Single-center, Randomized, Blinded, Placebo- and Active-controlled Crossover Study to Evaluate the Effect of Saroglitazar Magnesium on the QTc Interval in Healthy Volunteers
Brief Title: A Study to Evaluate the Effect of Saroglitazar Magnesium on the QTc Interval in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zydus Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: SARO.17.006
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Healthy
MeSH Terms: interventions — saroglitazar; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Study Treatment 1 (Experimental): Saroglitazar magnesium 4 mg
  Interventions: Drug: Saroglitazar magnesium 4mg
- Study treatment 2 (Experimental): Saroglitazar magnesium 20 mg
  Interventions: Drug: Saroglitazar magnesium 20 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebos
- Active Control (Active Comparator): Moxifloxacin 400 mg
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: Saroglitazar magnesium 4mg — 1 tablet of 4 mg Saroglitazar magnesium; 4 tablets of placebo to be administered orally
  Other Names: not any
  Arms: Study Treatment 1
Drug: Placebos — 5 tablets of placebo to be administered orally
  Other Names: not any
  Arms: Placebo
Drug: Moxifloxacin 400mg — 1 tablet of 400 mg Moxifloxacin to be administered orally
  Other Names: not any
  Arms: Active Control
Drug: Saroglitazar magnesium 20 mg — 5 tablets of 4 mg Saroglitazar magnesium to be administered orally
  Other Names: not any
  Arms: Study treatment 2

SUMMARY:
A Single-center, Randomized, Blinded, Placebo- and Active-controlled Crossover Study to Evaluate the Effect of Saroglitazar Magnesium on the QTc Interval in Healthy Volunteers

DETAILED DESCRIPTION:
Primary Objective: This is a Phase 1, single-center, blinded (with respect to saroglitazar magnesium and placebo administration), randomized, placebo- and active-controlled, 4-period crossover study to investigate the effect of single therapeutic and supra-therapeutic (5×) doses of saroglitazar magnesium on the corrected QT (QTc) interval in healthy subjects in compliance with the current version of the International Council for Harmonisation E14 Guidelines.

After confirmation of eligibility, 52 subjects (at least 16 will be females) will be randomly assigned to 1 of 4 treatment sequences using a William's design prior to study treatment administration on Day 1 of Period 1. Randomized subjects will receive each of the 4 study treatments across the 4 treatment periods separated by at least a 7-day washout period.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated written informed consent prior to any study-specific procedures
2. Willing and able to comply with the study procedures, restrictions, and requirements.
3. At least (≥) 18 years of age and no more than (≤) 45 years of age a
4. Body mass index of 19.0 to 25.0 kg/m² (inclusive) with a body weight of 50 to 100 kg
5. non-smokers and must not drink alcohol (teetotal).
6. Subjects who, in the opinion of the Investigator, are healthy as determined by their pre-study medical history, physical examination, and 12-lead ECG, and clinical laboratory tests within the institutional normal range or judged as not clinically significant by the Investigator, including the following parameters: hematology, serum biochemistry, urinalysis, and serology.
7. Male subjects and female subjects of childbearing potential must practice highly effective contraception during the study and be willing and able to continue contraception for 90 days after their last administration of study treatment.
8. Systemic blood pressure with a systolic blood pressure of 100 to 140 mmHg and a diastolic blood pressure of 60 to 90 mmHg.

Exclusion Criteria:

1. History of cardiovascular disease (eg, hypertension, arrhythmia, heart failure, long QT syndrome, or other conditions/diseases causing prolongation of the QT/QTc interval), in the opinion of the Investigator.
2. A prolongation of the QT interval corrected for HR using Fridericia's correction (QTcF) interval (eg, repeated demonstration of a QTcF interval >450 msec) before study treatment administration.
3. Any clinically important abnormalities in the ECG at screening, check-in (Day -1), or predose on Day 1. This includes subjects with any of the following:

   1. PR interval >210 msec;
   2. QRS >110 msec; or
   3. HR <45 beats per minute (bpm) or >100 bpm.
4. A QRS and/or T-wave value that the Investigator judges to be unfavorable for consistently accurate QT measurements (eg, indistinct QRS onset, low amplitude T-wave, inverted or terminally-inverted T-wave, merged T/U-waves, indistinct T-wave offset, or prominent U-wave that affects QT measurement).
5. History of additional risk factors for Torsades de Pointes or the presence of a family history of short QT syndrome, long QT syndrome, sudden unexplained death at a young age (≤40 years), drowning or sudden infant death syndrome in a first degree relative (ie, biological parent, sibling, or child).
6. Use of medications in the 90 days before Day -1 of Period 1 that are known to prolong the QT/QTc interval.
7. Has used prescription drugs and other substances (eg, dietary or herbal supplements such as St John's Wort) known to be either significant enzyme inducers or enzyme inhibitors within 4 weeks of Day 1 of Period 1, or use of grapefruit or similar substances (Seville oranges or marmalade, grapefruit juice, grapefruit hybrids, pomelos, exotic citrus fruits or fruit juices) within 7 days of Day 1 of Period 1.
8. Has used prescription or over-the-counter medication, excluding routine vitamins but including megadose vitamin therapy (intake of 20 to 600 times the recommended daily dose), within 7 days of Day 1 of Period 1, unless agreed as not clinically relevant by the Investigator and Sponsor.
9. Any history of malignant disease, including solid tumors, hematologic malignancies, and including any carcinoma in situ.
10. Clinically significant allergies, as determined by the Investigator.
11. History of any clinically significant endocrine, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major diseases, as determined by the Investigator.
12. History of unexplained syncopal or hypotensive episodes.
13. A positive cotinine test and positive breath test at screening or check-in (Day -1) of Period 1.
14. Surgery within 12 months prior to check-in (Day -1) of Period 1 (other than minor cosmetic surgery and minor dental surgery).
15. Subjects who have recent illness (eg, fever >38°C) within 7 days of check-in (Day -1) of Period 1.
16. Clinically significant abnormal hematology and serum biochemistry values, as determined by the Investigator or any of the following values at screening or check-in (Day -1) of Period 1:

    1. Alanine aminotransferase, aspartate aminotransferase, or creatinine above their reference range.
    2. Hemoglobin or platelets below their reference range.
17. Subjects with an absolute neutrophil count <2.0 × 10³/μL at screening or check-in (Day -1) of Period 1, any documented laboratory value <1.5 × 10³/μL, or any documented history of neutropenia.
18. Subjects with an estimated glomerular filtration rate (as defined by estimation of creatinine clearance using the Modification of Diet in Renal Disease formula) of ≤80 mL/min/1.73m² at screening.
19. History of, or positive screening test for, hepatitis C infection (defined as positive for hepatitis C virus antibody), hepatitis B infection (defined as positive for hepatitis B surface antigen), or human immunodeficiency virus I or II.
20. Treatment with saroglitazar magnesium, or any other PPAR agonist within 90 days prior to Day -1 of Period 1.
21. Treatment with another investigational drug or approved therapy for investigational use within 90 days of Day -1 of Period 1 or 5 × the t1/2 (whichever is longer), or the subjects is in follow-up for any other drug, biologic, or device study.
22. Current active infection or serious infection (eg, pneumonia, septicemia) within the 90 days prior to Day -1 of Period 1 as determined by the Investigator.
23. Female subjects who are pregnant, currently breastfeeding, or attempting to conceive.
24. Known hypersensitivity to either saroglitazar magnesium or other PPAR agonists, and or the excipients in the saroglitazar magnesium tablet formulation.
25. Known hypersensitivity to moxifloxacin or other quinolones.
26. Blood donation in the past 90 days, or bone marrow or stem cell donor in the past 12 months prior to check-in (Day -1) of Period 1.
27. Any disorder that, in the Investigator's opinion, may interfere with study compliance, such as significant mental, nervous disorder or other illness. In making this assessment, the Investigator must refer to the study information provided including the Investigator's Brochure, and the prescribing information for saroglitazar magnesium.
28. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol.
29. Inability to be venipunctured or tolerate venous puncture.
30. Any condition or abnormal baseline findings that in the Investigator's judgment might increase the risk to the subject or decrease the chance of obtaining satisfactory data needed to obtain the objective of the study.
31. Has acute gastrointestinal symptoms at the time of screening or check-in (Day -1) of Period 1 (eg, nausea, vomiting, diarrhea, heartburn).
32. Other unspecified reasons that, in the opinion of the Investigator or the Sponsor, make the subject unsuitable for the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2019-11-27 (Actual); Study Completion 2019-12-02 (Actual)

PRIMARY OUTCOMES:
QTcF change-from-baseline | Pre-dose (-1.0 hr) to 24 hours post dose
  Linear-mixed model will be used to assess the effect of saroglitazar magnesium on cardiac repolarization on Day 1 to evaluate whether saroglitazar magnesium prolongs the QTcF when orally administered to healthy volunteers
Saroglitazar and its metabolite saroglitazar sulfoxide plasma concentrations and placebo-corrected change-from-baseline QTcF | Pre-dose (-1.0 hr) to 24 hours post dose
  Quantification of the relationship between saroglitazar and its metabolite saroglitazar sulfoxide plasma concentrations and QTcF, using concentration-effect modeling

SECONDARY OUTCOMES:
Observed and change-from-baseline HR, PR, RR, QRS, and QT and ECG morphological abnormalities | Pre-dose (-1.0 hr) to 24 hours post dose
  Evaluation of the effect of Saroglitazar magnesium on other ECG parameters (ventricular HR, PR, RR, QRS, QT) and ECG morphological abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Deven V Parmar, MD,FCP, Study Director — Zydus Therapeutics Inc.
Locations (1):
- Cliantha Research Limited, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No